CLINICAL TRIAL: NCT07084961
Title: A Pharmacodynamic Study of TS-172 in Healthy Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TS172-03-09
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Healthy Adult Male Subjects

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TS-172 20 mg (sequence A) (Experimental)
  Interventions: Drug: TS-172
- TS-172 20 mg (sequence B) (Experimental)
  Interventions: Drug: TS-172

INTERVENTIONS:
Drug: TS-172 — Oral administration of TS-172 20 mg immediately before meal
Drug: TS-172 — Oral administration of TS-172 20 mg immediately after meal

SUMMARY:
An open-label, single-center, crossover study to evaluate the impact of administration timing of TS-172 on the pharmacodynamics in healthy adult male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Japanese healthy adult males whose age is >=18 and <40 years at the time of obtaining informed consent
2. Subjects whose body mass index is >=18.5 and <25.0 at the screening test
3. Subjects who are judged by a principal investigator or a sub-investigator to be eligible for participation in the study based on the results at the screening test and before administration of the drugs used in the study
4. Subjects who have been informed of the clinical trial, understand the details of the trial, and give their written consent prior to participation in the trial

Exclusion Criteria:

1. Subjects with medical history ineligible for participation in the study such as of respiratory, cardiovascular, gastrointestinal, hepatic, renal, urologic, endocrine, metabolic, hematologic, immunologic, dermatologic, neurologic, or psychiatric diseases
2. Subjects with medical history of disease (e.g., stomach or intestinal ulcers) or surgery (e.g., gastrectomy, gastric bandage, gastric bypass) that may affect the absorption of the drugs used in the study
3. Subjects who have been hospitalized with any treatment or undergone surgery within 12 weeks prior to receiving the drugs used in the study
4. Subjects with medical history of drug allergies (limited to severe symptoms such as anaphylaxis) or significant allergic predispositions (e.g., asthma that requires treatment)
5. Subjects who have used medications (including over-the-counter drugs) within 2 weeks prior to receiving the drugs used in the study

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2025-08-05 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
Urinaly excretion of phosphorus | Up to 3 days postdose during each period
Urinaly excretion of sodium | Up to 3 days postdose during each period

CONTACTS AND LOCATIONS:
Overall Officials: Taisho Director Taisho Director, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No